CLINICAL TRIAL: NCT02303795
Title: A Phase 2, Randomized, Open Label, Non-Inferiority Clinical Trial to Explore the Safety and Efficacy of Rivaroxaban Compared With Vitamin K Antagonism in Patients With Atrial Fibrillation With Bioprosthetic Mitral Valves - RIVER
Brief Title: RIvaroxaban for Valvular Heart diseasE and atRial Fibrillation Trial -RIVER Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIVER01
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Valvular Heart Disease
Keywords: bioprosthetic mitral valve; valvular heart disease; anticoagulant agents; NOACs; rivaroxaban; warfarin
MeSH Terms: conditions — Heart Valve Diseases | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban 20mg (Active Comparator): Oral Rivaroxaban, 20 mg od. Patients with a calculated creatinine clearance of 30 to 49 mL/min per 1.73 m2 received a reduced dose of rivaroxaban of 15 mg od.
  Interventions: Drug: Rivaroxaban; Drug: Warfarin
- Warfarin (Active Comparator): Warfarin Warfarin once daily (q.d.). The individual doses will be titrated as needed to maintain a target INR of 2.0-3.0.
  Interventions: Drug: Rivaroxaban; Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Patients assigned to rivaroxaban will receive oral rivaroxaban, 20 mg od. Patients with a calculated creatinine clearance of 30 to 49 mL/min per 1.73 m2 received a reduced dose of rivaroxaban of 15 mg od.
Drug: Warfarin — Patients will take the warfarin once daily (q.d.). The individual doses will be titrated as needed to maintain a target INR of 2.0-3.0.
  Patients with 65 > years old, should take warfarin (2,5mg/day) and all others patients should take 5mg/day.

SUMMARY:
RIvaroxaban for Valvular heart diseasE and atRial fibrillation trial (RIVER trial).

DETAILED DESCRIPTION:
A Phase 2, Randomized, Open label, Non-Inferiority Clinical Trial to Explore the Safety and Efficacy of Rivaroxaban compared with vitamin K antagonism in Patients with Atrial Fibrillation with Bioprosthetic Mitral valves - RIVER. Main analysis for the primary endpoint are based on the Restricted Mean Survival Time (RMST) method.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged >18 years at time of inclusion
2. Patients with Persistent or paroxysmal Atrial Fibrillation or flutter with bioprosthetic mitral valves.

   * The patient must be able to give informed consent

Exclusion Criteria:

1. Cardiovascular-related conditions as known presence of cardiac thrombus or tumor

   * Active endocarditis
   * Uncontrolled hypertension
2. Hemorrhage risk-related criteria

   * Active internal bleeding
   * History of, or condition associated with, increased bleeding risk
3. Concomitant conditions and therapies

   * History of previous thromboembolism with high risk of bleeding:

     * Severe, disabling stroke (modified Rankin score of 4-5, inclusive) within 3 months
     * Acute thromboembolic events or thrombosis (venous/arterial) within the last 14 days prior to randomization
     * Acute MI within the last 14 days prior to randomization
   * Treatment with: Chronic aspirin therapy > 100 mg daily or dual antiplatelet therapy; Intravenous antiplatelets; Fibrinolytics; Anticipated need for long-term treatment with a nonsteroidal antiinflammatory drug; Systemic treatment with a strong inhibitor of cytochrome P450 3A4, such as ketoconazole or protease inhibitors; Treatment with a strong inducer of cytochrome P450 3A4, such as rifampicin, phenytoin, phenobarbital, or carbamazepine.
   * Anemia
   * Pregnancy or breastfeeding or women of reproductive age not using effective contraceptive methods
   * Calculated creatinine clearance bellow 30 mL/min
   * Known significant liver disease or alanine aminotransferase N3× the upper limit of normal
   * Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Major Clinical Events | 12 months
  Combined Endpoint of major clinical events as defined by strokes (CVA), transient ischemic attack (TIA), major bleeding, all-cause death, valve thrombosis and non-CNS systemic embolism, hospitalization due to cardiac failure.

SECONDARY OUTCOMES:
Major bleeding | 12 months
  Clinically overt bleeding associated with: fatal outcome, involving a critical site, or clinically overt bleeding associated with a fall in hemoglobin concentration of ≥2 g/dL, or leading to transfusion of ≥2 units of packed red blood cells or whole blood.
Combined endpoint of nonfatal stroke (CVA), transient ischemic attack (TIA), systemic embolism, valve thrombosis, venous thromboembolism and vascular causes death.thrombosis, and vascular death | 12 months
  Stroke: sudden, focal neurologic deficit from a presumed cerebrovascular cause, not reversible within 24 hours and not due to na identifiable cause.
  Non-CNS systemic embolism: abrupt vascular insufficiency associated with clinical or radiologic evidence of arterial occlusion.
  Valve thrombosis: any thrombus attached to or near an implanted valve that occludes part of the blood flow, interferes with function or warrant treatment.
  Mortality: Deaths any cause. Venous thromboembolism: verification by definitive diagnostic evaluation. Deep Vein Thrombosis: abnormal compression ultrasound or intraluminal filling defect on venography or autopsy.
  Pulmonary embolism: at least one: 1) intraluminal filling defect on CT scan; 2) intraluminal filling defect on pulmonary angiogram; 3) high- probability on v/p lung scan; 4)inconclusive spiral CT, pulmonary image with demonstration of DVT in the lower extremities; 5) autopsy

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Berwanger, MD, PhD, Study Chair — Hospital do Coracao; Ricardo Pavanello, MD, PhD, Study Chair — Hospital do Coracao; Helio P Guimarães, MD, PhD, Principal Investigator — Hospital do Coracao
Locations (1):
- Associação do Sanatório Sírio - Hospital do Coração HCor, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Guimaraes HP, Lopes RD, de Barros E Silva PGM, Liporace IL, Sampaio RO, Tarasoutchi F, Hoffmann-Filho CR, de Lemos Soares Patriota R, Leiria TLL, Lamprea D, Precoma DB, Atik FA, Silveira FS, Farias FR, Barreto DO, Almeida AP, Zilli AC, de Souza Neto JD, Cavalcante MA, Figueira FAMS, Kojima FCS, Damiani L, Santos RHN, Valeis N, Campos VB, Saraiva JFK, Fonseca FH, Pinto IM, Magalhaes CC, Ferreira JFM, Alexander JH, Pavanello R, Cavalcanti AB, Berwanger O; RIVER Trial Investigators. Rivaroxaban in Patients with Atrial Fibrillation and a Bioprosthetic Mitral Valve. N Engl J Med. 2020 Nov 26;383(22):2117-2126. doi: 10.1056/NEJMoa2029603. Epub 2020 Nov 14. PMID 33196155
- [Derived] Guimaraes HP, de Barros E Silva PGM, Liporace IL, Sampaio RO, Tarasoutchi F, Paixao M, Hoffmann-Filho CR, Patriota R, Leiria TLL, Lamprea D, Precoma DB, Atik FA, Silveira FS, Farias FR, Barreto DO, Almeida AP, Zilli AC, de Souza Neto JD, Cavalcante MA, Figueira FAMS, Junior RA, Moises VA, Mesas CE, Ardito RV, Kalil PSA, Paiva MSMO, Maldonado JGA, de Lima CEB, D'Oliveira Vieira R, Laranjeira L, Kojima F, Damiani L, Nakagawa RH, Dos Santos JRY, Sampaio BS, Campos VB, Saraiva JFK, Fonseca FH, Pinto IM, Magalhaes CC, Ferreira JFM, Lopes RD, Pavanello R, Cavalcanti AB, Berwanger O; RIVER (RIvaroxaban for Valvular Heart diseasE and atRial Fibrillation Trial -RIVER Trial) Investigators. A randomized clinical trial to evaluate the efficacy and safety of rivaroxaban in patients with bioprosthetic mitral valve and atrial fibrillation or flutter: Rationale and design of the RIVER trial. Am Heart J. 2021 Jan;231:128-136. doi: 10.1016/j.ahj.2020.10.001. Epub 2020 Oct 10. PMID 33045224